CLINICAL TRIAL: NCT05034276
Title: Digital Therapeutic Development of Virtual Cognitive-Affective Training for Opioid Use Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: BehaVR LLC (Industry); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Eric Garland, Distinguished Professor, University of Utah
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB_00141495; R44DA053848 (NIH)
Record Dates: First submitted 2021-09-01; First posted 2021-09-05 (Actual); Results first posted 2023-07-20 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Opioid-use Disorder
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MORE-VR (Experimental): Mindfulness-Oriented Recovery Enhancement deployed over virtual reality.
  Interventions: Other: MORE-VR

INTERVENTIONS:
Other: MORE-VR — Mindfulness-Oriented Recovery Enhancement therapy delivered over virtual reality.

SUMMARY:
This is a Phase 1 trial that aims to establish the safety of MORE-VR, as well as to collect feasibility, usability, and engagement data, for patients receiving medications for opioid use disorder (mOUD).

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* DSM-5 opioid use disorder diagnosis
* treated with medications for opioid use disorder (MOUD)

Exclusion Criteria:

* Mindfulness intervention experience (MBSR, MBRP)
* Active psychosis or high risk of suicidality
* Cognitive impairment (per self-report or report by clinician)
* Unwilling or unable to remain in MOUD treatment for duration of study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2021-10-04 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-07-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Center on Mindfulness and Integrative Health Intervention Development, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Garland EL, Recasens M, Taple BJ, Donaldson GW, Weisberg RB. Virtual reality-based Mindfulness-Oriented Recovery Enhancement (MORE-VR) as an adjunct to medications for opioid use disorder: a Phase 1 trial. Ann Med. 2024 Dec;56(1):2392870. doi: 10.1080/07853890.2024.2392870. Epub 2024 Aug 22. PMID 39172534

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 34 participants were enrolled but only 28 participants started the intervention and attended the first treatment session. The other 6 participants were lost-to-follow up prior to initiation of the study intervention. This type of dropout is common among patients with opioid use disorder.
Period: Overall Study
Arm/Group | MORE-VR
Started | 28
Completed | 23
Not Completed | 5

BASELINE CHARACTERISTICS:
Arm/Group | MORE-VR
Number analyzed (Participants) | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.5 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 22
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 0
  White | 26
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 28

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events and/or Serious Adverse Events
Description: Number of participants who reported adverse events and serious adverse events.
Time Frame: Baseline through week 8
Measure: Count of Participants; unit: Participants
Arm/Group | MORE-VR
Number analyzed (Participants) | 28
Participants | 2

2. Secondary Outcome: Engagement
Description: Net Promoter Score (NPS) is a engagement and satisfaction measurement taken from asking participants how likely they were to recommend the MORE-VR intervention to others on a scale of 0-10. Net Promoter Score (NPS) is calculated by subtracting the percentage of customers who answer the NPS question with a 6 or lower (known as 'detractors') from the percentage of customers who answer with a 9 or 10 (known as 'promoters'). The summary Net Promoter Score is reflected as a percentage.
Time Frame: Baseline through week 8
Measure: Count of Participants; unit: Participants
Arm/Group | MORE-VR
Number analyzed (Participants) | 28
Participants | 20

3. Secondary Outcome: Numeric Rating Scale of State Craving
Description: Craving measured on a 0 to 10 numeric rating scale, with 0 indicating no craving and 10 indicating extreme craving.
Time Frame: Baseline through week 8
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | MORE-VR
Number analyzed (Participants) | 28
score on a scale | 1.22 (.23)

4. Secondary Outcome: Numeric Rating Scale of State Positive Affect
Description: Positive affect measured on a 0 to 10 numeric rating scale, with 0 indicating no positive affect and 10 indicating very high positive affect.
Time Frame: Baseline through week 8
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | MORE-VR
Number analyzed (Participants) | 28
score on a scale | 1.23 (.17)

5. Other Pre Specified Outcome: Desire for Drugs
Description: Desires for Drugs Questionnaire
Time Frame: Baseline, week 8
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Trait Positive and Negative Affect
Description: Positive and Negative Affect Schedule
Time Frame: Baseline, week 8
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Coping Self-efficacy
Description: Drug Taking Confidence Questionnaire
Time Frame: Baseline, week 8
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Cue-elicited Heart Rate
Description: Heart rate during cue exposure minus baseline heart rate
Time Frame: Baseline through week 8
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | MORE-VR
All-Cause Mortality (participants affected / at risk) | 0/28
Serious Adverse Events (participants affected / at risk) | 0/28
Other Adverse Events (participants affected / at risk) | 2/28
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MORE-VR (N=28)
Nausea (Gastrointestinal disorders) | 1 (1)
Panic attack (Psychiatric disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
This study was nonrandomized and cannot determine the efficacy of the intervention.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-09): https://cdn.clinicaltrials.gov/large-docs/76/NCT05034276/Prot_SAP_000.pdf